CLINICAL TRIAL: NCT03654976
Title: A Phase III Trial Evaluating the Efficacy and Safety of the House Dust Mite (HDM) Sublingual Immunotherapy (SLIT)-Tablet in Children and Adolescents (5-17 Years) With HDM Allergic Asthma
Brief Title: Mite Asthma Pediatric Immunotherapy Trial
Acronym: MAPIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-11; 2016-004363-39 (EudraCT Number)
Record Dates: First submitted 2018-08-24; First posted 2018-08-31 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Allergic Asthma Due to Dermatophagoides Farinae; Allergic Asthma Due to Dermatophagoides Pteronyssinus; Allergic Rhinitis Due to House Dust Mite
Keywords: Allergic asthma, allergic rhinitis, HDM, pediatric
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Subject's ICS or ICS/LABA background medication plus HDM SLIT-tablet
  Interventions: Biological: HDM SLIT-tablet
- Placebo (Placebo Comparator): Subject's ICS or ICS/LABA background medication plus placebo oral tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HDM SLIT-tablet — Sublingual allergy immunotherapy tablet, for daily administration (1 tablet per day)
  Other Names: Acarizax; Odactra
  Arms: Active treatment
Other: Placebo — Placebo sublingual tablet, for daily administration (1 tablet per day)
  Arms: Placebo

SUMMARY:
The trial aims to demonstrate efficacy of the House Dust Mite SLIT-tablet versus placebo as add-on treatment in children and adolescents (5-17 years) with House Dust Mite allergic asthma based on clinically relevant asthma worsening.

DETAILED DESCRIPTION:
The trial aims to demonstrate efficacy of the HDM SLIT-tablet versus placebo as add-on treatment in children and adolescents (5-17 years) with HDM allergic asthma based on clinically relevant asthma exacerbations.

Additionally, the trial will investigate if the treatment has an effect on asthma symptoms including nightly awakenings due to asthma, asthma medication use, asthma control, lung function, allergic rhinitis and allergic rhinoconjunctivitis.

Finally, quality of life (QoL) for subjects and caregivers will be measured.

The trial is a randomised, parallel-group, double-blind, placebo-controlled multi-national phase III trial conducted in Europe and North America. The treatment period will be approximately 2 years. Subjects will receive a written asthma action plan.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or female of any race/ethnicity aged 5-17 years
* A female subject of childbearing potential must have a negative pregnancy test and be willing to practise appropriate contraceptive methods
* A clinical history of HDM allergic asthma
* Use of low daily dose of ICS plus LABA or medium/high daily dose of ICS with or without LABA for the control of asthma symptoms
* A clinical history of asthma exacerbations in the past two years
* One or more of the following within the past 4 weeks prior to randomisation:

  * Daytime asthma symptoms more than twice/week
  * Any nocturnal awakening due to asthma
  * SABA rescue medication needed for treatment of asthma symptoms
  * Any activity limitation due to asthma
* Lung function measured by FEV1 ≥ 70% of predicted value or according to local requirements
* Clinical history of HDM AR within the last year prior to randomisation
* An average TCRS>0 during the baseline period
* Positive specific IgE (defined as ≥class 2, ≥0.70 kU/l) against D. pteronyssinus and/or D. farinae at screening
* Positive SPT to D. pteronyssinus and/or D. farinae at screening
* Subject willing and able to comply with trial protocol

Exclusion Criteria:

* Is sensitised and regularly exposed to animal dander, molds, and/or cockroach or other perennial allergen
* Has experienced a life-threatening asthma attack
* Within the last month before the randomisation visit (visit 3), has had an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalisation, or treatment with systemic corticosteroids
* Within the last 3 months before the randomisation visit (visit 3) while on high dose ICS treatment, has had an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalisation, or treatment with systemic corticosteroids
* Any SLIT or SCIT treatment with D. pteronyssinus or D. farinae within the previous 12 months
* Ongoing treatment with any allergy immunotherapy product
* Any clinically relevant condition or chronic disease incl. malignancy that in the opinion of the investigator would interfere with the trial evaluations or the safety of the subject
* Has a diagnosis of eosinophilic oesophagitis
* A relevant history of systemic allergic reactions
* Ongoing treatment with OCS
* Treatment with restricted and prohibited concomitant medication
* Treatment with an investigational drug within 30 days/5 half-lives of the drug (which ever longest) prior to screening
* A history of allergy, hypersensitivity or intolerance to any of the excipients or active substance of the IMP (except D. pteronyssinus and D. farinae) or to any excipient of the rescue medication provided in this trial
* A business or personal relationship with trial staff or sponsor who is directly involved with the conduct of the trial
* A history of alcohol or drug abuse
* Has previously been randomised into this trial, is participating in this trial at another investigational site or is participating or planning to participate in any other clinical trial during the duration of this trial
* Has a history or current evidence of any condition, treatment, laboratory values out of range or other circumstance that in the opinion of the investigator are clinically relevant and might expose the subject to risk by participating in the trial, confound the results of the trial, or interfere with the subject's participation for the full duration of the trial
* Has a condition or treatment that increase the risk of the subject developing severe adverse reactions after adrenaline/epinephrine administration
* Is unable to or will not comply with the use of adrenaline/epinephrine auto-injectors for countries where this is a regulatory requirement

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 533 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Roberts, MD, Principal Investigator — University Hospital Southampton NHS Foundation
Locations (64):
- United States (7):
  - Miami Clinical Research, Miami, Florida
  - Columbus Regional Research Institute, Columbus, Georgia
  - Respiratory Medicine Research Institute of MI, Ypsilanti, Michigan
  - Private Clinic, Bangor, Pennsylvania
  - Allergy Consultants, Verona, Pennsylvania
  - TTS research, Boerne, Texas
  - STAAMP Research, San Antonio, Texas
- Bulgaria (8):
  - MHAT, Plovdiv
  - UMBAL "St. Georgy", Plovdiv
  - SHATPPD, Rousse
  - Medical Center-1-Sevlievo EOOD, Sevlievo
  - Alitera-Med-Medical Center EOOD, Sofia
  - MBAL Tokuda Hospital Sofia, Sofia
  - Medical Center Excelsior, Sofia
  - DCC Ritam 2010, Stara Zagora
- France (5):
  - Hopital Augustin Morvan, Brest
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre hospitalier intercommunal, Créteil
  - Hôpital Jeanne de Flandre, Lille
  - Groupe hospitalier Armand Trousseau - La Roche Guyon, Paris
- Germany (3):
  - Kinderarzt-Praxis Bramsche, Bramsche
  - Kinderarztpraxis Ludwigsfelde, Ludwigsfelde
  - Kinderarztpraxis, Wuppertal
- Hungary (6):
  - Bajai Szent Rókus Kórház, Baja
  - Heim Pal Children's Hospital, Budapest
  - Semmelweis Egyetem, Budapest
  - Kanizsai Dorottya Korhaz, Nagykanizsa
  - Szent István Rendelő és Patika, Ráckeve
  - Aranyklinika Kft, Szeged
- Poland (15):
  - NZOZ E-Vita, Bialystok
  - Prywatna Praktyka Lekarska Gabinet Pediatryczno-Alergologiczny, Bialystok
  - Specjalistyczna Praktyka Lekarska, Katowice
  - Centrum Medyczne PROMED, Krakow
  - Centrum Nowoczesnych Terapii, Krakow
  - WWCOiT, Lodz
  - ALERGOTEST s.c. Specjalistyczne Centrum Medyczne, Lublin
  - Uniwersytecki Szpital Dzieciecy w Lublinie, Lublin
  - Ostrowieckie Centrum Medyczne S.C., Ostrowiec Świętokrzyski
  - Prywatny Gabinet Lekarski, Rzeszów
  - NSZOZ Puls, Skarżysko-Kamienna
  - ETG Skierniewice, Skierniewice
  - ALERGO-MED Specjalistyczna, Tarnów
  - Dobrostan, Wroclaw
  - Specjalist., Zabrze
- Russia (11):
  - Kazan State Medical University 138, Kazan'
  - First Moscow State Medical University, Moscow
  - Clinical and Diagnostic Centre "Zdorovie", Rostov-on-Don
  - Rayzan Regional Children Hospital, Ryazan
  - City children's polyclinic #35, Saint Petersburg
  - GBUZ "Children Municipal Polyclinic #45", Saint Petersburg
  - LLC ArsVite Severo-Zapad, Saint Petersburg
  - LLC Kurator, Saint Petersburg
  - GBUZ "Samarskiy oblastnoy detskiy sanatoriy "Yunost" 9-proseka, Samara
  - LLC 'ArsVitae Samara', Samara
  - Siberian State Medical University, Tomsk
- Spain (7):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital de Sagunto, Sagunto
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital de Conxo, Santiago de Compostela
  - Hospital de la Plana, Villarreal
- United Kingdom (2):
  - Royal Manchester Children's Hospital - Paediatrics Oxford Road, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts G, Just J, Nolte H, Hels OH, Emeryk A, Vidal C. SQ House Dust Mite Sublingual Immunotherapy Tablet in Children With Allergic Asthma: A Randomised Phase III Trial. Allergy. 2025 Dec;80(12):3401-3411. doi: 10.1111/all.70073. Epub 2025 Oct 9. PMID 41064908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial had randomized participants from 64 sites in 9 countries (Bulgaria, France, Germany, Hungary, Poland, Russia, Spain, United Kingdom, US).
Groups:
- HDM SLIT-tablet (12 SQ-HDM): Participant's daily background asthma medication of low dose inhaled corticosteroid (ICS) plus long-acting beta-agonist (LABA) or medium/high dose ICS with or without LABA, reliever asthma medication of short-acting beta-agonist (SABA) as needed plus 1 daily house dust mite (HDM) sublingual allergy immunotherapy tablet (12 SQ-HDM)
- Placebo SLIT-tablet: Participant's daily background asthma medication of low dose ICS plus LABA or medium/high dose ICS with or without LABA, reliever asthma medication of SABA as needed plus 1 daily placebo sublingual tablet
Period: Overall Study
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Started | 270 | 263
Completed IMP | 239 | 242
Full Analysis Set | 264 | 260
Safety Analysis Set | 270 | 263
Completed (Completed trial) | 241 | 245
Not Completed | 29 | 18
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Reason stated as 'Other' in CRF | 10 | 6
Not completed — Adverse Event | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- HDM SLIT-tablet (12 SQ-HDM): Participant's daily background asthma medication of low dose ICS plus LABA or medium/high dose ICS with or without LABA, reliever asthma medication of SABA as needed plus 1 daily HDM sublingual allergy immunotherapy tablet (12 SQ-HDM)
- Total: Total of all reporting groups
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet | Total
Number analyzed (Participants) | 270 | 263 | 533
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 270 | 263 | 533
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (3.4) | 10.6 (3.3) | 10.6 (3.4)
Age, Customized [Count of Participants; unit: Participants]
  Children (5-11 years) | 162 | 154 | 316
  Adolescents (12-17 years) | 108 | 109 | 217
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 94 | 182
  Male | 182 | 169 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 25 | 44
  Not Hispanic or Latino | 238 | 224 | 462
  Unknown or Not Reported | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 6 | 5 | 11
  White | 259 | 254 | 513
  Asian | 1 | 0 | 1
  Other | 4 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Bulgaria | 32 | 33 | 65
  France | 13 | 12 | 25
  Germany | 6 | 5 | 11
  Hungary | 18 | 19 | 37
  Poland | 146 | 145 | 291
  Russia | 19 | 19 | 38
  Spain | 20 | 16 | 36
  United Kingdom | 2 | 2 | 4
  United States | 14 | 12 | 26
Region [Count of Participants; unit: Participants]
  West (DEU, ESP, FRA, GRB, USA) | 55 | 47 | 102
  Central (POL) | 146 | 145 | 291
  East (BGR, HUN, RUS) | 69 | 71 | 140

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Clinically Relevant Asthma Exacerbations
Description: The primary endpoint of the trial was the annualized rate of clinically relevant asthma exacerbations calculated as the number of exacerbations per year per participant during the efficacy evaluation period of 20 months. A clinically relevant asthma exacerbation had to be medically confirmed and was defined as asthma worsening leading to at least 1 of the following criteria:
  * Doubling of ICS dose compared to background treatment
  * Systemic corticosteroids for treatment of asthma symptoms for at least 3 days
  * Emergency room visit due to asthma, requiring systemic corticosteroids
  * Hospitalization for more than 12 hours due to asthma, requiring treatment with systemic corticosteroids
  The outcome measure (by treatment group) is an adjusted annualized rate of clinically relevant asthma exacerbations.
Time Frame: Efficacy assessment period was 20 months (following a 4-10 months treatment initiation and maintenance period)
Population: Participant from the full analysis set with observations in the efficacy assessment period.
Measure: Mean (95% Confidence Interval); unit: Exacerbations per year per participant
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 252 | 257
Exacerbations per year per participant | 0.18 [0.13 to 0.25] | 0.21 [0.15 to 0.28]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The number of clinically relevant asthma exacerbations was analyzed using a negative binomial regression model with a log-link function and the logarithm of the time in years in the efficacy period as offset. The model included treatment, age group (<12 years, >=12 years) and region (west: DEU, ESP, FRA, GBR and USA; central: POL; east: BGR, HUN and RUS) as fixed factors. No missing data approach was applied; Test type: Superiority; p = 0.5412, Negative binomial regression; Rate ratio = 0.89, 95% CI 2-sided [0.60 to 1.31] — 12 SQ-HDM SLIT-tablet as the numerator and placebo SLIT-tablet as the denominator

2. Secondary Outcome: Proportion of Days With Nocturnal Awakenings Due to Asthma Requiring SABA Rescue Medication
Description: The days with nocturnal awakenings due to asthma requiring SABA rescue medication were entered in an eDiary by the participant/caregiver in a 2-week period every 4 months. The proportion of days with nocturnal awakenings due to asthma requiring SABA was presented on a range from 0 to 1 (1 indicating that all days in the eDiary period were with nocturnal awakenings due to asthma requiring SABA rescue medication). The efficacy assessment was based on data collected over the 20 months efficacy assessment period.
  The outcome measure (by treatment group) is an estimated proportion of days with nocturnal awakenings due to asthma requiring SABA rescue medication.
Time Frame: Efficacy assessment period was 20 months (following a 4-10 months treatment initiation and maintenance period)
Population: Participants from the full analysis set with observations in the efficacy assessment period.
Measure: Mean (95% Confidence Interval); unit: Proportion of days with awakenings
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 253 | 259
Proportion of days with awakenings | 0.0147 [0.0093 to 0.0233] | 0.0190 [0.0126 to 0.0287]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; A marginal logistic regression model with a generalized estimating approach was analyzed using treatment, visit, treatment*visit, age group (<12 years, >=12 years) and region (west: DEU, ESP, FRA, GBR and USA; central: POL; east: BGR, HUN and RUS) as fixed factors. Baseline visit was included as a covariate. No missing data approach was applied; Test type: Superiority; p = 0.4156, Marginal logistic regression; Odds Ratio (OR) = 0.7713, 95% CI 2-sided [0.41 to 1.44] — 12 SQ-HDM SLIT-tablet as the numerator and placebo SLIT-tablet as the denominator

3. Secondary Outcome: Proportions of Days With SABA Use
Description: The days with SABA use were entered in an eDiary by the participant/caregiver in a 2-week period every 4 months. The proportion of days with SABA use was presented on a range from 0 to 1 (1 indicating that all days in the eDiary period were with SABA use). The efficacy assessment was based on data collected over the 20 months efficacy assessment period.
  The outcome measure (by treatment group) is an estimated proportion of days with SABA use.
Time Frame: Efficacy assessment period was 20 months (following a 4-10 months treatment initiation and maintenance period)
Population: Participants from the full analysis set with observations in the efficacy assessment period.
Measure: Mean (95% Confidence Interval); unit: Proportion of days with SABA use
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 253 | 259
Proportion of days with SABA use | 0.0943 [0.0694 to 0.1269] | 0.1094 [0.0855 to 0.1391]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; A marginal logistic regression model with a generalized estimating approach was analyzed using treatment, visit, treatment*visit, age group (<12 years, >=12 years) and region (west: DEU, ESP, FRA, GBR and USA; central: POL; east: BGR, HUN and RUS) as fixed factors. Baseline visit is included as a covariate. No missing data approach was applied; Test type: Superiority; p = 0.4146, Marginal logistic regression; Odds Ratio (OR) = 0.8477, 95% CI 2-sided [0.57 to 1.26] — 12 SQ-HDM SLIT-tablet as the numerator and placebo SLIT-tablet as the denominator

4. Secondary Outcome: Percentage Predicted FEV1
Description: The outcome measure (by treatment) is an average of the percentage predicted FEV1 measured at visits 5 to 11 (every 4 months during the 20 months efficacy assessment period), analyzed using MMRM (mixed-effect model repeated measurement).
  FEV1 (forced expired volume in 1 second) is assessed by use of spirometry and is a measure for lung function. Percentage predicted FEV1 is derived from the predicted FEV1, which is the expected value of FEV1 for a person of a certain age, race, height and gender with healthy lungs.
Time Frame: Efficacy assessment period was 20 months (following a 4-10 months treatment initiation and maintenance period)
Population: Participants from the full analysis set with observations in the efficacy assessment period
Measure: Mean (95% Confidence Interval); unit: Percentage predicted FEV1
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 254 | 259
Percentage predicted FEV1 | 97.17 [96.02 to 98.32] | 97.05 [95.82 to 98.28]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; A 'mixed-effect model repeated measurement' model was analysed using treatment, visit, treatment*visit, age group (<12 years, >=12 years) and region (west: DEU, ESP, FRA, GBR and USA; central: POL; east: BGR, HUN and RUS) as fixed factors. Baseline visit was included as a covariate. No missing data approach was applied; Test type: Superiority; p = 0.8829, Mixed-effect model repeated measurement; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-1.47 to 1.70] — 12 SQ-HDM - placebo

5. Secondary Outcome: Global Evaluation of Allergic Asthma as Having an Improved Outcome
Description: At the end of trial visit, the subject was asked, when compared to their asthma before IMP treatment, how they felt overall. Subjects who answered 'much better' or 'better' were categorized as having improved allergic asthma. At the end of trial visit, subjects had been treated for 24-30 months (including a 4-10 months treatment initiation and maintenance period).
  The outcome measure (by treatment) is an adjusted odds of experiencing improved allergic asthma.
Time Frame: Assessment done at the end of trial visit (after 24-30 months of treatment)
Population: Participants from the full analysis set with observations in the efficacy assessment period
Measure: Mean (95% Confidence Interval); unit: Odds of improved allergic asthma
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 239 | 244
Odds of improved allergic asthma | 14.66 [8.30 to 25.89] | 6.48 [4.03 to 10.43]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The odds of having an improved outcome was analyzed using a generalized linear mixed model (GLMM) with a logit link function. The model included treatment, age group (<12 years, >=12 years) and region (west: DEU, ESP, FRA, GBR and USA; central: POL; east: BGR, HUN and RUS) as fixed factors. No missing data approach was applied; Test type: Superiority; p = 0.0044, Generalised linear mixed model; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.29 to 3.96] — 12 SQ-HDM SLIT-tablet as the numerator and placebo SLIT-tablet as the denominator

6. Secondary Outcome: Global Evaluation of Allergic Rhinitis as Having an Improved Outcome
Description: At the end of trial visit, the subject was asked, when compared to their rhinitis before IMP treatment, how they felt overall. Subjects who answered 'much better' or 'better' were categorized as having improved allergic rhinitis. At the end of trial visit, subjects had been treated for 24-30 months (including a 4-10 months treatment initiation and maintenance period).
  The outcome measure (by treatment) is an adjusted odds of experiencing improved allergic rhinitis.
Time Frame: Assessment done at the end of trial visit (after 24-30 months of treatment)
Population: Participants from the full analysis set with observations in the efficacy assessment period.
Measure: Mean (95% Confidence Interval); unit: Odds of improved allergic rhinitis
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
Number analyzed (Participants) | 239 | 244
Odds of improved allergic rhinitis | 8.29 [5.35 to 12.85] | 5.11 [3.49 to 7.48]
Statistical Analysis 1: Comparison: HDM SLIT-tablet (12 SQ-HDM) vs Placebo SLIT-tablet; The odds of having an improved outcome was analysed using a generalised linear mixed model (GLMM) with a logit link function. The model included treatment, age group (<12 years, >=12 years) and region (west: DEU, ESP, FRA, GBR and USA; central: POL; east: BGR, HUN and RUS) as fixed factors. No missing data approach was applied; Test type: Superiority; p = 0.0698, Generalised linear mixed model; Odds Ratio, log = 1.62, 95% CI 2-sided [0.96 to 2.74] — 12 SQ-HDM SLIT-tablet as the numerator and placebo SLIT-tablet as the denominator

7. Other Pre Specified Outcome: Allergic Rhinitis Symptoms
Description: Allergic rhinitis symptoms were entered in an eDiary by the participant/caregiver in a 2-week period every 4 months, for up to 24-30 months.
Time Frame: The efficacy assessment period for the endpoint started 4 months after treatment initiation and lasted until the end of the trial or discontinuation of treatment (up to 24-30 months of treatment).
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Allergic Rhinitis Medication Use
Description: Allergic rhinitis medication use were entered in an eDiary by the participant/caregiver in a 2-week period every 4 months, for up to 24-30 months.
Time Frame: as for outcome 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs were collected from consent to last follow-up phone contact (up to 24-30 months of treatment).
Description: Treatment emergent AEs (TEAEs) are displayed (these were AEs starting on/after time of first IMP and no later than 7 days after last day of IMP). For the first 28 days of treatment, the presence/absence of 15 specific symptoms, identified as local side effects of sublingual immunotherapy (solicited events), were captured in an eDiary. Solicited events were evaluated by the investigator and reported in the eCRF as AEs as per their discretion. TEAEs from the eCRF are included in TEAEs presented.
Groups:
- Placebo SLIT-tablet: Participant's daily background asthma medication of low dose ICS plus LABA or medium/high dose ICS with or without LABA, reliever asthma medication of SABA as needed plus 1 daily placebo sublingual allergy immunotherapy tablet
Arm/Group | HDM SLIT-tablet (12 SQ-HDM) | Placebo SLIT-tablet
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/263
Serious Adverse Events (participants affected / at risk) | 14/270 | 12/263
Other Adverse Events (participants affected / at risk) | 250/270 | 228/263
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDM SLIT-tablet (12 SQ-HDM) (N=270) | Placebo SLIT-tablet (N=263)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Testicular cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HDM SLIT-tablet (12 SQ-HDM) (N=270) | Placebo SLIT-tablet (N=263)
Ear pruritus (Ear and labyrinth disorders) | 104 (257) | 60 (124)
Conjunctivitis allergic (Eye disorders) | 14 (19) | 12 (13)
Abdominal pain upper (Gastrointestinal disorders) | 118 (231) | 101 (194)
Aphthous ulcer (Gastrointestinal disorders) | 16 (28) | 17 (28)
Diarrhoea (Gastrointestinal disorders) | 60 (96) | 51 (77)
Glossodynia (Gastrointestinal disorders) | 74 (134) | 18 (23)
Lip swelling (Gastrointestinal disorders) | 71 (154) | 14 (18)
Mouth swelling (Gastrointestinal disorders) | 67 (159) | 11 (16)
Mouth ulceration (Gastrointestinal disorders) | 26 (44) | 16 (17)
Nausea (Gastrointestinal disorders) | 85 (167) | 57 (96)
Oral pruritus (Gastrointestinal disorders) | 175 (475) | 65 (126)
Swollen tongue (Gastrointestinal disorders) | 55 (98) | 8 (8)
Tongue ulceration (Gastrointestinal disorders) | 19 (34) | 9 (15)
Vomiting (Gastrointestinal disorders) | 33 (49) | 14 (19)
Corona virus infection (Infections and infestations) | 18 (18) | 14 (14)
Nasopharyngitis (Infections and infestations) | 63 (110) | 57 (95)
Pharyngitis (Infections and infestations) | 21 (28) | 15 (21)
Upper respiratory tract infection (Infections and infestations) | 26 (38) | 25 (31)
Viral infection (Infections and infestations) | 18 (18) | 18 (22)
Dysgeusia (Nervous system disorders) | 54 (120) | 44 (68)
Headache (Nervous system disorders) | 16 (17) | 11 (13)
Asthma (Respiratory, thoracic and mediastinal disorders) | 80 (158) | 96 (176)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 20 (24)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 58 (113) | 14 (23)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 16 (27) | 23 (47)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 166 (494) | 94 (178)
Pyrexia (General disorders) | 12 (14) | 17 (19)
Bronchitis (Infections and infestations) | 12 (17) | 21 (29)
Influenza (Infections and infestations) | 12 (14) | 14 (16)

LIMITATIONS AND CAVEATS:
Enrollment was paused at the outbreak of the COVID-19 pandemic. During the COVID-19 pandemic the asthma exacerbation rate decreased both in the trial population (blinded data) and in the general asthma population. It was therefore deemed difficult to recruit participants based on a history of recent asthma exacerbations. The sponsor decided to end the trial with the completed participants on 10-Aug-2022 due to the severe impact of COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall be able to review any proposed publication or presentation at least 60 days in advance of submission. Sponsor cannot require changes. Upon sponsor's request, the investigator shall delay a publication or presentation for 6 months to permit the sponsor to take necessary steps to protect confidential information. For this multi-site trial it is mandatory that the primary publication is based on data from all trial sites analyzed as stipulated in the protocol and in the SAP.

DOCUMENTS (2):
  • Study Protocol (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT03654976/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT03654976/SAP_001.pdf